CLINICAL TRIAL: NCT02147093
Title: CLARITI (TM) 1-Day Multifocal Contact Lenses Performance and Acceptance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5175
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-06

CONDITIONS: Presbyopia Correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (sphere) /Test (multi-focal) (Other): Subjects were first fitted with Control lens (sphere) and a pair of reading glasses for one week. Subjects were then fitted with the Test lens (multi-focal) for one week.
  Interventions: Device: Test (multi-focal); Device: Control (Sphere)
- Test (sphere) /Control (multi-focal) (Other): Subjects were first fitted with the Test lens (multi-focal) for one week. Subjects were then fitted with Control lens (sphere) and a pair of reading glasses for one week.
  Interventions: Device: Test (multi-focal); Device: Control (Sphere)

INTERVENTIONS:
Device: Test (multi-focal) — contact lens was to be worn a daily wear.
  Other Names: Clariti 1 Day; filcon II 3
Device: Control (Sphere) — contact lens was to be worn a daily wear with spectacles
  Other Names: filcon II 3

SUMMARY:
A comparative evaluation of a newly marketed multifocal contact lens with a single vision contact lens when used with near vision spectacles. The evaluation was to quantify the difference between the two test corrections.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 years or more
2. Spectacle or soft contact lens wearer
3. Refraction: best sphere (corrected for back vertex distance) -6.00 Diopters (D) to +4.00 D; Astigmatism - 0.00 D to -0.75 D; Near addition for 40 cm; Medium Add: +1.50 D to +2.00 D; High Add: +2.25 D to +2.50 D
4. Best spectacle corrected visual acuity of 6/9 or better in each eye
5. Willingness to adhere to the instructions set forth in the clinical protocol
6. Signature of the subject Informed Consent form after review of Information to Participant document.

Exclusion Criteria:

1. Systemic or ocular allergies which might interfere with contact lens wear
2. Systemic disease which might interfere with contact lens wear
3. Ocular disease which might interfere with contact lens wear (e.g. hypothesia, insufficient lacrimal secretion)
4. Use of medication which might interfere with contact lens wear
5. Active ocular infection
6. Use of ocular medication
7. Significant ocular anomaly
8. Presence of two or more corneal scars in either eye
9. Monovision contact lens wearers
10. Pregnancy or lactation
11. Any medical condition that might be prejudicial to the study
12. Participants non-able to give consent or from a vulnerable group
13. Infectious disease (for example, hepatitis, tuberculosis, etc.) or a contagious immunosuppressive disease (such as HIV, AIDS, etc.)
14. Employees or family member of the investigational clinic (e.g. investigator, coordinator, technician)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 subjects were enrolled in this study. Of the enrolled subjects 1 did not meet the eligibility criteria and 40 subjects were dispensed a study lens. Of the dispensed subjects, 3 were discontinued and 37 subjects completed the study.
Groups:
- Control (Filcon II 3- Sphere) /Test (Filcon II 3-multi-focal): Subjects were first fitted with the Control lens (filcon II 3- sphere) and a pair of reading glasses for one week. Subjects were then fitted with the Test lens (filcon II 3-multi-focal) for one week.
- Test (Filcon II 3-multi-focal) /Control (Filcon II 3- Sphere): Subjects were first fitted with the Test lens (filcon II 3-multi-focal) for one week. Subjects were then fitted with Control lens (filcon II 3- sphere) and a pair of reading glasses for one week.
Period: Period 1
Arm/Group | Control (Filcon II 3- Sphere) /Test (Filcon II 3-multi-focal) | Test (Filcon II 3-multi-focal) /Control (Filcon II 3- Sphere)
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2
Arm/Group | Control (Filcon II 3- Sphere) /Test (Filcon II 3-multi-focal) | Test (Filcon II 3-multi-focal) /Control (Filcon II 3- Sphere)
Started | 20 | 19
Completed | 18 | 19
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were randomized to one of two lens wear serquences.
Groups:
- Control (Filcon II 3-sphere) /Test (Filcon II 3-multi-focal); Test (Filcon II 3-multi-focal) / Control (Filcon II 3-spher): All subjects that were randomized to sequence and were dispensed a study lens.
- Total: Total of all reporting groups
Arm/Group | Control (Filcon II 3-sphere) /Test (Filcon II 3-multi-focal) | Test (Filcon II 3-multi-focal) / Control (Filcon II 3-spher) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.20 (7.682) | 58.00 (9.067) | 56.78 (8.490)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Distance LogMAR Visual Acuity
Description: Distance time controlled LogMAR (Logarithm of the Minimum Angle of Resolution) Visual Acuity was carried out binocularly, at 4m (meter) under 250 cd/m^2 and 2.5 cd/m^2 (candela per square meter) luminance. The test was presented under the two conditions; High luminance (250 cd/m^2) High Contrast (90%) & Low Contrast (10%) and Low Luminance (2.5 cd/m^2) High Contrast (90%)
Time Frame: 7 days post wear
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Control (Filcon II 3-sphere): Subjects that were dispensed the Control lens (filcon II 3-sphere) in either the first or second period of the study.
- Test (Filcon II 3-multi-focal): Subjects that were dispensed the Test lens (filcon II 3-multi-focal) in either the first or second period of the study.
Arm/Group | Control (Filcon II 3-sphere) | Test (Filcon II 3-multi-focal)
Number analyzed (Participants) | 37 | 37
LogMAR
  High Contrast-Distance-Standard High Luminance | -0.466 (0.9995) | -0.972 (1.0104)
  Low Contrast-Distance-Standard High Luminance | -2.842 (1.6850) | -3.768 (1.8023)
  High Contrast-Distance-Standard Low Luminance | -2.834 (1.0042) | -3.700 (0.8939)

2. Primary Outcome: Near LogMAR Visual Acuity
Description: Near time controlled LogMAR Visual Acuity was carried out binocularly, at 4cm under 250 cd/m^2 and 50 cd/m^2 luminance. The test was presented on under the two conditions; High Luminance (250cd/m^2) High Contrast (90%) & Low Contrast (10%) and Low Luminance (50cd/m^2) High Contrast (90%)
Time Frame: 7 days post wear
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Control (Filcon II 3-sphere) | Test (Filcon II 3-multi-focal)
Number analyzed (Participants) | 37 | 37
LogMAR
  High Contrast-Near-Standard High Luminance | -1.455 (0.6309) | -2.545 (1.1240)
  Low Contrast-Near-Standard High Luminance | -2.151 (1.0221) | -3.820 (1.4124)
  High Contrast-Near-Standard Low Luminance | -1.878 (1.0546) | -3.441 (1.3941)

ADVERSE EVENTS:
Time Frame: Throughout duration of the study(approximately 4 months).
Arm/Group | Control (Filcon II 3-sphere) | Test (Filcon II 3-multi-focal)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days